CLINICAL TRIAL: NCT07389447
Title: FUS of the Dentate Nucleus and Superior Cerebellar Peduncle of the Cerebellum Induces Changes to EEG Power Bands, Spatiotemporal Dynamics, and Cognitive Function in Healthy Humans
Brief Title: Focused Ultrasound Stimulation of the Cerebellum to Induce Changes in Cognition and Brain Activity
Acronym: FUSCBM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Mohammad Alkhawashki, Dr, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: F1298R
Record Dates: First submitted 2025-08-06; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Trauma; Cognition; Agency; Verbal Memory; CCAS
Keywords: Cerebellum; Focused Ultrasound; Brain Stimulation; Computational Neuroscience; Neuroinformatics; White Matter; Grey Matter; Dentate Nucleus; Superior Cerebellar Peduncle; EEG; Power Band; Dynamics
MeSH Terms: conditions — Stroke; Wounds and Injuries | interventions — Electroencephalography

STUDY DESIGN:
Intervention Model Description: Participants will receive a sham and two target stimulations in different orders.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham (Sham Comparator): FUS transducer is off, otherwise the process is the same
  Interventions: Procedure: Focused ultrasound; Diagnostic Test: EEG
- Dentate (Active Comparator): FUS parameters set to target dentate with pre-specified distance and intensity
  Interventions: Procedure: Focused ultrasound; Diagnostic Test: EEG
- Superior cerebellar peduncle (Active Comparator): FUS parameters set to target superior cerebellar peduncle with pre-specified distance and intensity
  Interventions: Procedure: Focused ultrasound; Diagnostic Test: EEG

INTERVENTIONS:
Procedure: Focused ultrasound — Focused ultrasound stimulation administered to the cerebellar nucleus or efferent fiber tract.
  Other Names: FUS; tFUS; LIFUS
Diagnostic Test: EEG — This is the electroencephalography reading that will show changes in brain activity as describes in outcome measures

SUMMARY:
The goal of this preclinical study is to assess the effects of focused ultrasound stimulation to the cerebellum on brain dynamics and cognition in healthy volunteers aged 18 to 40. The main questions it aims to answer are:

Does FUS applied to the cerebellum affect cognition?

Does FUS applied to the white matter or gray matter of the cerebellum with the same parameters result in different outcomes?

Researchers will compare active and sham stimulations.

Participants will be asked to complete cognitive tasks after receiving FUS to the cerebellum.

ELIGIBILITY:
Exclusion Criteria:

* Participants must not have claustrophobia or anxiety regarding MRI scan.
* Participants must not have current or planned pregnancy.
* Participants must not have history of neurological or psychiatric disorder.
* Participants must not have predisposition for fainting spells (syncope).
* Participants must not have implanted material (e.g., pacemaker, neurostimulator, medication infusion device, cochlear implants).
* Participants must not have medical patch that cannot or may not be taken off (e.g., nicotine patch).
* Participants must not be currently taking psychoactive medication, or must have stopped taking such medication for at least 2 weeks before starting experiment (excluding contraception).
* Participants must not have skin disease on or close to the scalp.
* Participants must not have direct relatives (parents, siblings, children) with epilepsy, convulsion, or seizure.
* Participants must abstain from the use of any recreational drugs in the 48-hour period prior to taking part in the experiment.
* Participants must not consume more than 4 alcoholic units within the 24-hour period before participation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram (EEG) power and spatiotemporal dynamics | Through study completion, peri-procedurally, on days 1, 2 and 3
  The investigators measure the changes in EEG power in delta, theta, alpha, beta and gamma band, and spatiotemporal dynamics while administering concurrent transcranial focused ultrasound stimulation (tFUS). The EEG will also be used to asses network changes during sonication.
Electrooculogram (EOG) power and spatiotemporal dynamics | Through study completion, peri-procedurally, on days 1, 2 and 3
  The investigators measure the ocular saccades from both frontal head electrodes and electrodes places by the sides of the eyes while administering concurrent tFUS. This data will be used for identifying and removing eye-movement artifacts from EEG and assess eye saccades during sonication. This will be applied to some of the participants but not all, due to availability.

SECONDARY OUTCOMES:
Brief Ataxia Rating Scale (BARS) | Through study completion, post-procedurally, on days 1, 2 and 3
  The investigators measure BARS out of a total score of 30. A score of 0 means that the participant experiences no motor deficits of cerebellar origin, whereas a score of 30 means that the participant is highly ataxic.
Cerebellar Cognitive Affective Syndrome Scale (CCASS) | Through study completion, post-procedurally, on days 1, 2 and 3
  The investigators measure CCASS out of a total score of 120, or an absolute score that isn't limited, where a higher score is a better outcome
n-Back Continuous performance task | Through study completion, post-procedurally, on days 1, 2 and 3
  The investigators measure working memory with a game that involves remembering the last letter shown, with the "n" in n-Back denoting how many letters back the memorised letter was shown.
Agency Task | Through study completion, post-procedurally, on days 1, 2 and 3
  The investigators measure participant's sense of agency through a game which involves the participant assessing their level of control and performance. the score is calculated from how well the participant matches their assessment to the game's assessment.
Verbal Paired Associates (VPA) | Through study completion, post-procedurally, on days 1, 2 and 3
  The investigators measure a participant's ability to remember the second word in a set of word pairs. The score is out of a total of 48, but calculations are done to assess performance over repetitions and time.

OTHER OUTCOMES:
Heart rate | Through study completion, pre-procedurally, on days 1, 2 and 3
  Heart rate is measured to take a baseline reading prior to sonication. A stable heart rate between 60 and 80 bpm is favorable. A heart rate above 100 bpm or a low heart rate under 50 prompts us to reassess participant readiness. Heart rate is taken again post sonication only in case of adverse reaction.
Subjective experience | Through study completion, post-procedurally, on days 1, 2 and 3
  The participants will be questioned on their experience of the study and on any side effects they experience during or 24 hours after the stimulation. This isn't a scale but a questionnaire that has multiple measures such as sleepiness prior to experiment, and self reporting on adverse effects like dizziness or any other effects.
Blood Pressure | Through study completion, pre-procedurally, on days 1, 2 and 3
  Blood pressure is taken prior to sonication for baseline reading. A favorable reading falls within the normal range of 100/60 to 130/90. anything that falls outside of that range prompts reassessment of participant readiness. Blood pressure readings are taken again in case of any adverse reaction only.

CONTACTS AND LOCATIONS:
Locations (1):
- Precision Medical Imaging, QMC, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code